CLINICAL TRIAL: NCT07317115
Title: Magnetic Compression Anastomosis in Side-to-Side Duodeno-ileostomy Versus Semaglutide in Adults With Obesity and Type 2 Diabetes (MAGvMED Study)
Brief Title: Side-to-Side Duodeno-ileostomy Versus Semaglutide in Adults With Obesity and Type 2 Diabetes
Acronym: MAGvMED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GT Metabolic Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GTM-021
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Obesity (Disorder); Obesity & Overweight; Type 2 Diabetes (T2DM)
Keywords: Magnet System; Semaglutide; GT Metabolic Solutions, Inc.
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: 1:1 randomization of Surgery (MagDI System) versus Medication (semaglutide). At Day 360, subjects in the Medication arm will have the option to crossover to the Surgery Arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery Arm (Active Comparator): Magnet System
  Interventions: Device: Magnet System
- Medication Arm (Active Comparator): Semaglutide
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Device: Magnet System — Magnet System for side-to-side magnetic compression anastomosis in a duodeno-ileostomy bipartition
  Arms: Surgery Arm
Drug: Semaglutide — Semaglutide (up to 2.4mg subcutaneous (SQ) injection weekly or dose tolerated according to side effects); a glucagon-like peptide-1 receptor agonist (GLP-1RA)
  Arms: Medication Arm

SUMMARY:
Compare use of the Magnet System in side-to-side duodeno-ileostomy (Surgery) with semaglutide (Medication).

DETAILED DESCRIPTION:
Compare functional improvement of T2D using the Magnet System in duodeno-ileostomy for intestinal diversion versus semaglutide in eligible participants with obesity (BMI 30 - 40 kg/m2) and T2D (HbA1c ≥ 6.5%).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 30 - 40 kg/m2 and qualifies for obesity treatment at the discretion of the treating investigator (i.e., must be assessed to qualify for both surgery and medication treatment to justify randomization).
* Type 2 diabetes (T2D defined as HbA1c ≥ 6.5%).
* Participant agrees to refrain from additional metabolic and bariatric (MBS) or reconstructive surgery that would affect body weight for the duration of the study.
* Participant agrees to refrain from taking any additional semaglutide-containing or other GLP-1RA medication for the duration of the study, regardless of randomization assignment (i.e., Surgery or Medication).

Participant has been informed of the nature of the study and is willing and able to comply with requirements, including randomization, and provides written informed consent to participate in the study.

Exclusion Criteria:

* Meets any of the contraindications for either treatment arm (Surgery: Magnet System; or Medication: semaglutide), thereby prohibiting randomization
* Current or previous metabolic and bariatric surgery (MBS) treatment in the previous 12 months (e.g., sleeve gastrectomy, intragastric balloons, adjustable gastric banding).
* Taking or treated with semaglutide, semaglutide-containing medications, or any other GLP-1RA medication in the previous 12 months.
* Pregnant, lactating or planning pregnancy during the clinical study and follow-up period.
* Currently participating in an investigational drug, biologic, or medical device or other interventional clinical study.
* Presence of other anatomic or comorbid conditions, or medical, social or psychological conditions that, in the investigator's opinion, would contraindicate either treatment arm or could limit the participant's ability to participate in the clinical study or to comply with follow-up requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Functional improvement of T2D: HbA1c | Day 360

CONTACTS AND LOCATIONS:
Locations (1):
- Westmount Surgical Center, Westmount, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No